CLINICAL TRIAL: NCT06351748
Title: Real-world Study of CHina Ozempic cLinicAl pRactice in Patients With Type 2 Diabetes (SCHOLAR)
Acronym: SCHOLAR
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9535-7877; U1111-1296-3151 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with T2DM: Participants diagnosed with T2DM who initiated semaglutide OW for the first time between 1 Jan 2022 (the date when semaglutide OW was listed in the National Reimbursement Drug List [NRDL] in China) and 28 Feb 2023 (9 months prior to the data extraction cut-off date of 30 Nov 2023.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Participants received semaglutide OW according to local label and to routine clinical practice at the discretion of the treating physician.
  Other Names: Ozempic

SUMMARY:
This study is to describe the real-world use and impact of semaglutide once-weekly (OW) among participants with type 2 diabetes mellitus (T2DM) in China. Participants diagnosed with T2DM who initiated semaglutide OW for the first time between 1 Jan 2022 (the date when semaglutide OW was listed in the National Reimbursement Drug List [NRDL] in China] and 28 Feb 2023 (9 months prior to the data extraction cut-off date of 30 Nov 2023) will be included in this study. The study period will be 36 months prior to the first date of participants identification period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged greater than or equal to (≥) 18 years on index date
* Participants with diagnosis of T2DM prior to or on index date
* Participants with initiation of semaglutide OW for the first time within the identification period

Exclusion Criteria:

* Participants with diagnosis of type 1 diabetes prior to or on index date
* Participants who were pregnant within 36 months prior to or on index date
* Participants who participated in any clinical trials within 36 months prior to or on index date which could be identified from medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with T2DM who initiated semaglutide OW for the first time during the patient identification period.
Sampling Method: Probability Sample
Enrollment: 34238 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Change in Haemoglobin A1c (HbA1c) level | From baseline (3 months prior to or on the index date) to 6 months
  Measured in Percentage (%).
Change in HbA1c level | From baseline (3 months prior to or on the index date) to 6 months
  Measured in millimoles per mol (mmol/mol)
Proportion of participants achieving HbA1c less than (<) 7.0% | At 6 months
  Measured in percentage of participants.

SECONDARY OUTCOMES:
Change in HbA1c level | From baseline (3 months prior to or on the index date) to 12 months
  Measured in %.
Change in HbA1c level | From baseline (3 months prior to or on the index date) to 12 months
  Measured in mmol/mol.
Proportion of participants achieving HbA1c <7.0% | At 12 months
  Measured in percentage of participants.
Change in body weight | From baseline (3 months prior to or on the index date) to 12 months
  Measured in kilograms.
Change in body weight | From baseline (3 months prior to or on the index date) to 6 months
  Measured in kilograms.
Description of participants with different demographic characteristics | At baseline (12 months prior to or on the index date)
Description of participants with different clinical characteristics | At baseline (36 months prior to or on the index date)
Proportion of participants with different antidiabetic medications | At baseline (3 months prior to or on the index date)
  Measured in percentage of participants.
Proportion of participants with different non-antidiabetic medications | At baseline (3 months prior to or on the index date)
  Measured in percentage of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Tianjin Medical University Chu Hsien-I Memorial Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com